CLINICAL TRIAL: NCT05074537
Title: The WIIA - The Wright Center of Innovation Imaging Archive
Brief Title: The Wright Center of Innovation Imaging Archive
Acronym: WIIA
Status: Active, not recruiting | Type: Observational
Sponsor: University of Cincinnati (Other)
Responsible Party: Principal Investigator, Michael V Knopp MD PhD, Professor, University of Cincinnati
Other Study IDs: RP0310/2017H0429
Record Dates: First submitted 2019-11-25; First posted 2021-10-12 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Medical Imaging Data

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- MRI Participants
  Interventions: Diagnostic Test: MRI exam
- PET/CT Participants
  Interventions: Diagnostic Test: PET/CT imaging exam
- CT Participants
  Interventions: Diagnostic Test: CT imaging exam

INTERVENTIONS:
Diagnostic Test: MRI exam — Participants who are receiving standard of care or investigational MRI exams at the Wright Center will be eligible for enrollment in this data bank.
  Groups: MRI Participants
Diagnostic Test: PET/CT imaging exam — Participants who are receiving standard of care or investigational PET/CT exams at the Wright Center will be eligible for enrollment in this data bank.
  Groups: PET/CT Participants
Diagnostic Test: CT imaging exam — Participants who are receiving standard of care or investigational CT exams at the Wright Center will be eligible for enrollment in this data bank.
  Groups: CT Participants

SUMMARY:
This data bank will serve as a data resource for a multidisciplinary team of clinicians and basic scientists. Specifically, this data bank will allow investigators to generate preliminary data for competitive consideration in intermural and extramural funding while enabling advanced analytical tool development and deep learning methodologies. This effort will enable the use for leading edge innovation in biomedical imaging by using clinical imaging studies that otherwise could not be used for such developments. We aim to use these data to improve diagnostics and disease management. With this data bank, we hope to improve the quality of imaging and the precision of imaging based analytics to better detect potential health risks, predict treatment response, and monitor disease progression in order to guide management of future patients.

DETAILED DESCRIPTION:
The constant advances in computational capabilities and abilities of deep learning necessitate the availability of large imaging data sets that can be further analyzed. We therefore create the WIIA - The Wright Center of Innovation Imaging Archive - to serve as a repository for advanced data analytics and simulation. This will provide researchers access to a robust, comprehensive pool of imaging data for impactful research. The patient population under study includes adults who are 18 years of age and older. Children will be excluded from this study as they are unable to give voluntary consent. A partial waiver of HIPAA authorization will be requested to permit access to and use of PHI for recruitment purposes. However, investigational data will only be collected once consent to participate in the study is acquired. There will be no upper limit to the number of people who participate in this study. We expect 100-150 participants per year, with plans for the study to continue indefinitely. Data collected will include coded demographics, abbreviated medical history, current diagnoses, coded medical reports, coded surgical/nonsurgical treatment procedures, and follow up information. These data will be collected from Standard of Care (SOC) or investigational imaging studies. These data will be coded and stored in the Wright Center of Innovation Imaging Archive, which is a secure database of imaging studies. Data will be stored indefinitely. Administrative staff will construct and maintain the database as well as conduct annual quality assurance assessments of bank data. Oversight of the bank will be the responsibility of the Principal and Co-Investigators of the study. To maximize the use of this data bank and to promote collaborative, multi-institutional research, we are not limiting future data use. Data may be shared with Ohio State or non-Ohio State researchers. However, only investigators with sound, hypothesis driven research proposals can request data by completing a Data Request Form. This study will impose minimal medical risk to participants. At data leak is the primary risk, which will be minimized through precautions to protect PHI. Nevertheless, in the event of a data breach, the nature of the collected data ensures minimal financial or professional impact on the patient. This study does not confer a direct benefit to the patient. However, society may benefit from imaging advancements that arise from future studies using this data.

ELIGIBILITY:
Inclusion Criteria:

* Patient provides consent
* Patient is receiving or has received a SOC or investigational imaging scan

Exclusion Criteria:

* Patient does not wish to or is unable to provide consent
* Patient is below the age of 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patient population under study includes adults who are 18 years of age and older. Children will be excluded from this study as they are unable to give voluntary consent. A partial waiver of HIPAA authorization will be requested to permit access to and use of PHI for recruitment purposes. However, investigational data will only be collected once consent to participate in the study is acquired.
  Participants can include or donate their imaging data independently if it was performed at OSU or outside of OSU. For example, a subject may be willing to donate an imaging study performed previously or for different purposes and provides the WIIA with a CD or other data set.
  There will be no upper limit to the number of people who participate in this study. We expect 100-150 participants per year, with plans for the study to continue indefinitely.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2028-05 (Estimated); Study Completion 2030-05 (Estimated)

PRIMARY OUTCOMES:
Image quality | through study completion (roughly 10 years)
  We will be assessing image quality using a likert scale
Anatomic Variability - Likert Scale | through study completion (roughly 10 years)
Anatomic Variability - Length | through study completion (roughly 10 years)
Anatomic Variability - Volume | through study completion (roughly 10 years)
Anatomic Variability - Density | through study completion (roughly 10 years)

CONTACTS AND LOCATIONS:
Locations (1):
- Martha Morehouse Medical Plaza, Columbus, Ohio, United States

DOCUMENTS (1):
  • Study Protocol (2017-12-20): https://cdn.clinicaltrials.gov/large-docs/37/NCT05074537/Prot_000.pdf